CLINICAL TRIAL: NCT05468879
Title: Bioequivalence Study of 3 mg Glimepiride Tablet in Indonesia Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT Harsen Laboratories (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 540/STD/PML/2020
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Drug Use
Keywords: Bioequivalence study; Glimepiride; Indonesia; cross-over design study; pharmacokinetics
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Intervention Model Description: Randomized, single blind, two-period, single dose, cross-over study with one week washout period under fasted condition
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glimepiride 3 mg Tablet (Experimental): Participants received Glimepiride 3 mg Tablet with 240 mL of 20% glucose solution
  Interventions: Drug: Glimepiride
- Amaryl® 3 mg tablet (Active Comparator): Participants received Amaryl® 3 mg tablet (Glimepiride 3 mg) with 240 mL of 20% glucose solution
  Interventions: Drug: Amaryl®

INTERVENTIONS:
Drug: Glimepiride — Glimepiride is a sulfonylurea, indicated as an adjunct to proper dietary management, exercise and weight reduction to lower the blood glucose in patients with type 2 diabetes whose hyperglycemia cannot be controlled by diet and exercise alone.
  Arms: Glimepiride 3 mg Tablet
Drug: Amaryl® — Amaryl®
  Arms: Amaryl® 3 mg tablet

SUMMARY:
The study was conducted toinvestigate whether the bioavailability of 3 mg Glimepiride Tablet Manufactured by PT. Harsen Laboratories was bioequivalent to the reference product, 3 mg Amaryl® Tablet Manufactured by PT. Aventis Indonesia Pharma, Indonesia.

DETAILED DESCRIPTION:
The study was conducted following an oral administration of one tablet of the test drug (3 mg Glimepiride Tablet) or one tablet of the reference drug (3 mg Amaryl® Tablet ). Blood samples were drawn before dosing (0 h) and at 15, 30, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12, 18, 24, and 30 hours after drug administration. The entire subjects were given 60 mL of 20% glucose solution to minimize hypoglycemic effects at 15, 30, 45 minutes, and 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75 and 4 hours after drug administration. Following a washout period of one week, this procedure was repeated using the alternate drug. The plasma concentrations of glimepiride were determined by means of LC-MS/MS system. The LLOQ is 1.99 ng/mL of glimepiride. The pharmacokinetic parameters used in this study were area under the concentration-time curve of glimepiride from time zero to 30 hours (AUCt), area under the concentration-time curve from time zero to infinite (AUCinf), maximum concentration (Cmax), time required to reach the maximum concentration (tmax) and the elimination half life (t½).

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female
* had read the subject information and signed informed consent documents
* were age between 18 to 55 years
* had body mass index between 18 to 25 kg/m2
* had a normal electrocardiogram
* had normal blood pressure (systolic was ranged between 90 to 120 mmHg and diastolic was ranged between 60 to 80 mmHg)
* had normal heart rate (ranged between 60 to 100 bpm)
* have no significant disease in medical history; have no significant abnormal values in laboratory and physical examination during screening
* had acceptance to use protection (condom) during intercourse with their spouse throughout the study

Exclusion Criteria:

* Pregnant and/or nursing woman.
* Those with a history of contraindication or hypersensitivity to glimepiride, other antidiabetic agent or other ingredients in the study products or a history of serious allergic reaction to any drug, significant allergic disease or allergic reaction.
* Those with a history or presence of medical condition which might significantly influence the pharmacokinetics of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease.
* Those with a history or presence of any coagulation disorder or clinically significant hematology abnormalities.
* Those who using any medication (prescription or non-prescription drug, food supplement, herbal medicine), particularly the medication known to affect the pharmacokinetic of the study drug, within one week prior to the drug administration day.
* Those who had participated in any clinical study within 3 months prior to the study (< 90 days).
* Those who donated or lost 300 mL (or more) of blood within 3 months prior to the study.
* Those who smoked more than 10 cigarettes a day
* Those with a history of travelling to another city within the last 14 days
* Those with a history of direct contact with a COVID-19 positive person in the subject's neighborhood
* Those with a history or present of sore throat, fever (with temperature more than 37°C) or dyspnea within the last 14 days
* Those who reactive to anti SARS CoV-2 test
* Those who were positive to HIV, HBsAg, and HCV tests (to be kept confidential).
* Those with a history of drug or alcohol abused within 12 months prior to screening for this study
* Those who were unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | before dosing (0 hour) and at 15, 30, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12, 18, 24, and 30 hours after drug administration
  90% Confidence Interval
Area Under Curve from 0 to 30 hours (AUCt) | before dosing (0 hour) and at 15, 30, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12, 18, 24, and 30 hours after drug administration
  90% Confidence Interval

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | before dosing (0 hour) and at 15, 30, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12, 18, 24, and 30 hours after drug administration
  Pharmacokinetics Parameter
Area Under Curve from 0 to 30 hours (AUCt) | before dosing (0 hour) and at 15, 30, 45 minutes, and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 9, 12, 18, 24, and 30 hours after drug administration
  Pharmacokinetics Parameter

CONTACTS AND LOCATIONS:
Locations (1):
- PT Pharma Metric Labs, Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Liu Y, Zhang MQ, Zhu JM, Jia JY, Liu YM, Liu GY, Li S, Weng LP, Yu C. Bioequivalence and pharmacokinetic evaluation of two formulations of glimepiride 2 mg: a single-dose, randomized-sequence, open-label, two-way crossover study in healthy Chinese male volunteers. Clin Ther. 2010 May;32(5):986-95. doi: 10.1016/j.clinthera.2010.04.016. PMID 20685507
- [Background] Jung SH, Chae JW, Song BJ, Kwona KI. Bioequivalence Comparison of Two Formulations of Fixed-Dose Combination Glimepiride/Metformin (2/500 mg)Tablets in Healthy Volunteers. Iran J Pharm Res. 2014 Spring;13(2):365-71. PMID 25237332
- [Background] Zhu J, Li Y, Xiang Y, Zhou L, Li Y. Magnetic solid phase extraction followed with LC-MS/MS for determination of glimepiride in beagle dog plasma and its application to bioequivalence study. J Pharm Biomed Anal. 2020 May 30;184:113180. doi: 10.1016/j.jpba.2020.113180. Epub 2020 Feb 15. PMID 32092631
- [Result] Jovanovic D, Stojsic D, Zlatkovic M, Jovic-Stosic J, Jovanovic M. Bioequivalence assessment of the two brands of glimepiride tablets. Vojnosanit Pregl. 2006 Dec;63(12):1015-20. doi: 10.2298/vsp0612015j. PMID 17252706
- See also: Amaryl® (Glimepiride) Tablet 1,2, and 4 mg, Product Monograph — https://www.accessdata.fda.gov/drugsatfda_docs/label/2009/020496s021lbl.pdf